CLINICAL TRIAL: NCT02055014
Title: Randomisation to Endoluminal Intestinal Liner Alone Versus With Incretin Analogue in SustainEd Diabesity (REVISE-Diabesity)
Brief Title: Randomisation to Endobarrier Alone Versus With Incretin Analogue in SustainEd Diabesity (REVISE-Diabesity)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Collaborators: Association of British Clinical Diabetologists (Unknown)
Responsible Party: Principal Investigator, Dr Bob Ryder, Chief Investigator, Consultant Physician (Diabetes), Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12DIAB15; ISRCTN00151053 (Registry Identifier: ISRCTN); 2012-004988-42 (EudraCT Number)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes; Obesity; Diabesity
Keywords: Endobarrier; Duodenal-jejunal bypass liner; Glucagon-like peptide-1 receptor agonist; Liraglutide; Diabesity; Type 2 diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabesity | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Liraglutide alone (Active Comparator): Liraglutide 1.8mg once daily subcutaneous injection
  Interventions: Drug: Liraglutide
- Endobarrier alone (Experimental): Duodenal-jejunal bypass liner (Endobarrier) device implantation without additional GLP-1RA therapy
  Interventions: Device: Duodenal-jejunal bypass liner - Endobarrier device
- Endobarrier and Liraglutide (Experimental): Duodenal-jejunal bypass liner (Endobarrier) device with combined liraglutide 1.2mg once daily subcutaneous injection
  Interventions: Drug: Liraglutide; Device: Duodenal-jejunal bypass liner - Endobarrier device

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Endobarrier and Liraglutide; Liraglutide alone
Device: Duodenal-jejunal bypass liner - Endobarrier device
  Other Names: EC Certificate Full Quality Assurance System: Certificate US08/5323
  Arms: Endobarrier alone; Endobarrier and Liraglutide

SUMMARY:
New effective non-surgical treatments are needed for patients whose obesity and type 2 diabetes (T2DM) do not respond to current medical therapies. We propose a randomised controlled trial of Endobarrier, an implantable intestinal device that separates ingested food from contacting the first 60cm of intestine where sited and that mimics some of the clinical effects of bariatric surgery (improved metabolic control with weight loss) with or without continued use of the GLP-1 receptor agonist (GLP-1RA) Liraglutide 1.2mg vs Liraglutide 1.8mg without the device in obese patients with T2DM who remain with suboptimal glycaemic control despite current conventional diabetes treatment, in an NHS setting.

Seventy-two patients with T2DM and obesity (HbA1c≥7.5%, BMI≥35kg/m2) despite previous GLP-1RA therapy will be studied over 24 months and randomised to receive Endobarrier with continued Liraglutide 1.2mg for 12 months; Endobarrier alone for 12 months; or Liraglutide 1.8mg without Endobarrier.

We will investigate potential mechanisms of action and their time course as part of the study by repeated measures of: 1. insulin resistance measures, gut peptides, bile acids; 2. energy intake and nutritional composition; 3. liver fat stores, 4. intestinal inflammation and permeability measures.

The data will inform clinical use of the device and development of new treatments for T2DM and obesity.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes with latest HbA1c ≥7.5% (≥58mmol/mol)
* obesity with latest BMI ≥35 Kg/m2 (≥30 Kg/m2 for those of South Asian origin)
* liraglutide therapy for at least 6 months - HbA1c and weight trend data should be available
* stable weight and HbA1c in preceding 3 months (<3 Kg reduction in weight and <0.3% reduction in HbA1c)

Exclusion Criteria:

* <18 years of age
* abnormal intestinal anatomy e.g. Crohn's disease
* contraindication to oesophago-gastroduodenoscopy
* previous bariatric surgery or bowel surgery
* active infection
* anticoagulation therapy which cannot be discontinued/ coagulopathy INR >1.3
* eGFR <30
* known portal hypertension
* previous pancreatitis or amylase > 3 times the upper limit of normal
* uncontrolled cardiovascular disease
* lactating or pregnant females
* patients taking aspirin in whom it should continue (e.g. active ischaemic heart disease or cerebrovascular disease)
* excess anaesthetic risk as identified by the anaesthetist or investigator (e.g. uncontrolled obstructive sleep apnoea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | 24 months
  HbA1c (mmol/mol; %) at end of follow-up period compared to baseline. This will be 12 months following Endobarrier device removal which will usually be 24 months after initial the device has first been implanted (for 12 months) or 24 months from Liraglutide 1.8mg initiation.

SECONDARY OUTCOMES:
Weight | 24 months
  Weight (Kg) measured at end of follow-up period compared to baseline. This will be 12 months following Endobarrier device removal which will usually be 24 months after the device has first been implanted (for 12 months) or 24 months from Liraglutide 1.8mg initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Ryder, MD FRCP, Principal Investigator — Sandwell and West Birmingham Hospitals NHS Trust
Locations (4):
- United Kingdom (4):
  - Department of Diabetes, City Hospital, Birmingham
  - Glasgow Royal Infirmary, Glasgow
  - Department of Diabetes, Guy's and St Thomas' Hospitals, London
  - Diabetes Research Group, King's College London, London